CLINICAL TRIAL: NCT01201681
Title: Peri-operative Pain and Root Canal Therapy
Brief Title: DPBRN Peri-operative Pain and Root Canal Therapy
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other); University of Florida (Other); University of Copenhagen (Other); University of Alabama at Birmingham (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Gregg H. Gilbert, DDS, MBA, FAAHD, Professor and Chair, General Dental Sciences, Dental Practice-Based Research Network
Other Study IDs: 133266; U01DE016747 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Post-operative Tooth Pain; Root Canal Therapy
Keywords: Post-operative pain; intra-operative pain; root canal therapy; feasibility; post-surgical persistent pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post-operativeTooth Pain

SUMMARY:
The purpose of this study is to identify pre-operative factors that put patients at greater risk of developing severe tooth pain following root canal therapy, thereby providing evidence that will allow dentists to act preventively to lessen this risk, improve pain control, increase their patients' quality of life, and decrease the number of dental emergency interactions.

A parallel goal of this study is to assess the feasibility of recruiting dentists that provide root canal therapy and patients using the DPBRN.

DETAILED DESCRIPTION:
Goals for this study is to:

* Assess the frequency and intensity of pre-operative pain
* Evaluate the occurence and intensity of intra-operative pain
* Evaluate the occurence and intensity of post-operative pain
* Assess the interference of persistent tooth pain with daily life
* Identify a limited set of risk factors related to the development of post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* 19-70 years old
* permanent adult tooth requiring it first non-surgical root canal therapy
* patients with more than 1 tooth requiring root canal therapy are eligible, but only the first root canal procedure performed will be included to avoid problems of correlation within patients

Exclusion Criteria:

* Evidence of prior root canal therapy, including iatrogenic, but not disease-induced, pulp access of the tooth being considered
* patients with obvious cognitive impairments (e.g., past stroke with communication deficits, dementia, mental disability)
* patients unable to return for 6 month follow-up, since another study plans to obtain data of these patients at that time (DPBRN Persistent Tooth Pain)

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants directly involved in this study are patients who have sought dental treatment in the practitioner-investigators' practices. The practitioner-investigators will be endodontists and general dentists.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Nixdorf, DDS, MS, Principal Investigator — University of Minnesota
Locations (8):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida College of Dentistry, Gainesville, Florida
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon
- University of Copenhagen Royal Dental College, Copenhagen, Denmark

REFERENCES:
- [Derived] Nixdorf DR, Law AS, Lindquist K, Reams GJ, Cole E, Kanter K, Nguyen RHN, Harris DR; National Dental PBRN Collaborative Group. Frequency, impact, and predictors of persistent pain after root canal treatment: a national dental PBRN study. Pain. 2016 Jan;157(1):159-165. doi: 10.1097/j.pain.0000000000000343. PMID 26335907
- [Derived] Law AS, Nixdorf DR, Aguirre AM, Reams GJ, Tortomasi AJ, Manne BD, Harris DR; National Dental PBRN Collaborative Group. Predicting severe pain after root canal therapy in the National Dental PBRN. J Dent Res. 2015 Mar;94(3 Suppl):37S-43S. doi: 10.1177/0022034514555144. Epub 2014 Oct 29. PMID 25355775
- [Derived] Law AS, Nixdorf DR, Rabinowitz I, Reams GJ, Smith JA Jr, Torres AV, Harris DR; National Dental PBRN Collaborative Group. Root canal therapy reduces multiple dimensions of pain: a national dental practice-based research network study. J Endod. 2014 Nov;40(11):1738-45. doi: 10.1016/j.joen.2014.07.011. Epub 2014 Sep 1. PMID 25190605
- See also: Dental Practice-Based Research Network — http://DPBRN.org
- See also: Dental Practice-Based Research Network — http://DentalPBRN.org